CLINICAL TRIAL: NCT05398107
Title: Building Emotion Awareness and Mental Health (BEAM) Program for Mothers of Children 6-18 Months Old: A Pilot Randomized Control Trial and Community Partnership With Family Dynamics
Brief Title: Building Emotion Awareness and Mental Health (BEAM): Community Partnership With Family Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other); Tactica Interactive (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAM FD
Record Dates: First submitted 2022-04-26; First posted 2022-05-31 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-03

CONDITIONS: Depression, Anxiety
Keywords: Mental health; Parenting; Maternal; Psychoeducation; E-health; mhealth
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: This pilot Randomized Controlled Trial will involve two arms. Participants randomized to the BEAM program or the standard of care, MoodMission. The experimental arm will include 40 mothers in the BEAM program while the standard of care will include 40 mothers. Randomization will be stratified based on the telehealth group timeslots mothers are available for.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: The BEAM program (Experimental): The BEAM Program is delivered through a mobile application, weekly group telehealth sessions, and an online community forum. BEAM includes ~ 20 minutes of weekly video modules on parenting and mental health. Mental health videos provide content and emotion-regulation strategies drawn from the Unified Protocol, an evidence-based treatment for depression and anxiety disorders. Self-compassion and effective communication are also central focuses of the mental health content. Supportive parenting videos will provide mothers with emotion-focused parenting strategies and help mothers understand and respond to their children's challenging emotions and behaviours. The weekly group telehealth sessions will allow mothers to discuss content and ask questions, with the purpose of developing a sense of community and social support. The online community forum will provide a space for mothers to reflect on their learned skills and connect with other mothers taking part in the program.
  Interventions: Behavioral: Experimental: Building Emotion Awareness and Mental Health (BEAM)
- Standard of Care: MoodMission (Active Comparator): MoodMission is an evidence-based app which was developed based on cognitive behavioural therapy (CBT). The MoodMission app will provide mothers with missions. Missions are mental health strategies based on scientific evidence which are easily achievable (e.g., relaxation tips, exercise and fitness activities, yoga, mindfulness meditations, affirmations and coping statements). MoodMission will tailor missions based on the mothers current mood.
  Interventions: Behavioral: Control: MoodMission

INTERVENTIONS:
Behavioral: Experimental: Building Emotion Awareness and Mental Health (BEAM) — The BEAM Program is based on best-practices in telehealth and science-based program design aimed at promoting maternal mental health and supportive parenting. The BEAM Program app is hosted on the University of Manitoba secure servers and is designed/managed by Tactica Interactive. The weekly group telehealth sessions will be led by clinical coaches (a mental health professional or Doctoral-Level Clinical Psychology Student) and will use the secure videoconferencing platform Zoom (Healthcare license). Parent coaches will be mothers who have recently participated in a prior iteration of the BEAM program. Parent coaches will engage with participants on the community peer support forum and will also attend weekly telehealth sessions. The therapeutic aims of the BEAM program are to improve symptoms of anxiety and depression as well as parenting skills, and will emphasize self-compassion, effective communication practices, and social support networks.
  Arms: Experimental: The BEAM program
Behavioral: Control: MoodMission — MoodMission will be used as our Standard of Care control group. MoodMission is an app based on CBT principles which creates tailored "missions" for mothers. These missions are based on self-reported mood and are aimed to improve mental health symptoms.
  Arms: Standard of Care: MoodMission

SUMMARY:
Throughout the COVID-19 pandemic, postpartum depression and anxiety has increased dramatically. This is problematic as mothers in Manitoba must wait 12-18 months for therapeutic services. Children exposed to maternal mental illness in the first few years of life are at risk of negative lifelong adverse effects. Thus, the investigators of this project created and have tested The Building Emotion Awareness and Mental health (BEAM) program, which is an app-based mental health and parenting program for mothers of young children who are experiencing depression and/or anxiety. BEAM is now ready to be tested in partnership with an established community agency. This partnership will enable counsellors to provide expert-led mental health treatment to supplement and expand upon existing mental health services and will enable an established agency to address widespread unmet family mental health needs through the provision of mobile health (mHealth) content, training, and consultation. A two-arm pilot randomized controlled trial (RCT) with repeated measures will be used to evaluate the BEAM program compared to MoodMission (an evidence-based mHealth program) which will be the standard of care. Outcomes will be assessed to determine the effects of the BEAM program on reducing maternal mental health symptoms among a sample of 80 mothers who self-report moderate-to-severe symptoms of depression and/or anxiety (on the Patient Health Questionnaire-9 and the Generalized Anxiety Disorder-7, respectively), meet criteria for a current major depressive episode and/or anxiety disorder (as determined on the Mini International Neuropsychiatric Interview) and have a child between the ages of 6 to 18 months old.

DETAILED DESCRIPTION:
Maternal depression and anxiety levels have increased dramatically throughout the COVID-19 pandemic. Studies show as many as 25-30% of mothers are experiencing clinically significant symptoms. Children exposed to maternal depression early in life are more likely to experience irritable temperament, socio-emotional developmental impairments, sleep concerns, and are at a long-term risk of lifelong mental illness. Thus, given the high rate of young children born throughout the pandemic who were exposed to maternal depression and anxiety, there is a critical need to mitigate these potential negative impacts on young children. In Manitoba, there is a serious gap in mental health services, with mothers waiting upwards of 12-18 months for therapy on provincial waitlists. Typically, programs that address both child and mother mental health are effective. However, these programs are usually costly, require highly trained clinicians, and have lengthy waitlists. Mobile apps show promising results for treating depression and anxiety but are rarely targeted towards mothers. Many of these factors led the investigators of this project to create the Building Emotion Awareness and Mental health (BEAM) program, which is a mobile health (mHealth) program designed to mitigate the impacts of pandemic stress on family mental health and includes (1) expert-led psychoeducational and parenting strategies videos; (2) structured group sessions to enhance therapeutic content and build social supports; (3) a monitored online forum to enhance peer connection; and (4) symptom monitoring to track progress.

The pilot results for the BEAM program among mothers of infants has shown promising results. The investigators noted statistically significant reductions in depression, anxiety, parenting distress, and child internalizing symptoms following the intervention for BEAM participants versus participants in the standard of care. The investigators are now ready to partner with an established community agency, Family Dynamics, who will be provided with BEAM training and consultation. mHealth apps are usually delivered by third parties without involving trusted community agencies who have a sense of local needs and can offer additional supports if needed. Unfortunately, family agencies typically lack the infrastructure and personnel capacities to adequately treat maternal mental illness. The BEAM program will enable counsellors to provide expert-led mental health treatment which will supplement and expand upon existing services provided at Family Dynamics. This partnership approach with Family Dynamics will enable an established agency to address widespread unmet family mental health needs.

There are two primary aims to this study:

1. To determine the efficacy of BEAM compared to MoodMission, an app-based cognitive behavior therapy for treatment of moderate depression and anxiety, at reducing outcomes of interest in a randomized controlled trial (RCT). Primary (maternal depression and anxiety), secondary (maternal mental health, parenting, and child), and exploratory (relationship and weekly maternal mental health) outcomes will be assessed.
2. To examine the efficacy, feasibility, and acceptability of the BEAM program when delivered by a community agency, compared to MoodMission, while exploring opportunities for program development.

ELIGIBILITY:
Inclusion Criteria:

* Mother with a child 6 to 18 months old
* Moderate-to-severe symptoms of depression and/or anxiety (i.e., a score at or above 10 on the Patient Health Questionnaire and/or the General Anxiety Disorder scale)
* Comfortable understanding, speaking, and reading English
* Residing in the province of Manitoba, Canada
* Willing to complete pre-intervention, post-intervention, and follow-up questionnaires (approximately 45 minutes each)
* Willing to complete a one hour mental health interview with a trained student on the Mini International Neuropsychiatric Interview (MINI)
* Meets criteria for a major depressive episode or anxiety disorder (i.e., (i.e., panic disorder, agoraphobia, social anxiety disorder, post traumatic stress disorder, or generalized anxiety disorder)
* Availability to attend weekly telehealth sessions

Exclusion Criteria:

* Suicide attempt within the past year
* Self-harm in past 6 months
* Clinically significant psychotic symptoms on the MINI
* A diagnosis of post-traumatic stress disorder on the MINI which, in clinical opinion, would make it impossible for the mother to participate in the program
* A diagnosis of severe alcohol use disorder and/or a substance use disorder on the MINI which, in clinical opinion, would make it impossible for the mother to participate in the program
* Lives outside of Manitoba, Canada
* Does not meet criteria for moderate-to-severe depression and/or anxiety on the PHQ-9 and/or GAD-7
* Child is outside of the 6 to 18 month age range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in maternal depression | The PHQ-9 will be administered during the eligibility screening (up to 2 months before randomization), pre-intervention (T1), during the weekly surveys (up to 11 weeks), after the intervention (T2; after week 12), and at a 6-month follow-up (T3).
  Symptoms of depression will be assessed using the Patient Health Questionnaire-9. The Patient Health Questionnaire-9 is a self-administered questionnaire with possible scores ranging from 0 to 27, where higher scores are indicative of more severe symptoms. Data analyses will assess total Patient Health Questionnaire-9 scores as well as cut-off scores (≥ 10).
Changes in maternal anxiety | The GAD-7 will be completed during the eligibility screening (up to 2 months before randomization), pre-intervention (T1), during the weekly surveys (up to 11 weeks), after the intervention (T2; after week 12), and at a 6-month follow-up (T3).
  Symptoms of anxiety will be assessed using the Generalized Anxiety Disorder 7-Item scale. The Generalized Anxiety Disorder-7 Item is a self-administered questionnaire with possible scores ranging from 0 to 21, where higher scores are indicative of more severe symptoms. Data analyses will assess total Generalized Anxiety Disorder-7 Item scores as well as cut off scores (≥ 10).

SECONDARY OUTCOMES:
Changes in parenting stress | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2: 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Symptoms of parenting stress will be assessed using the Parenting Stress Index-Short Form, which has three subscales measuring parental distress, parent-child dysfunction, and difficult child. Scores can range from 15 to 100, with higher scores indicating higher stress levels. Data analyses will assess total Parenting Stress Index-Short Form and subscale scores.
Changes in maternal sleep disturbance | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Symptoms of sleep disturbance will be assessed using the sleep disturbance subscale of the Patient Reported Outcomes Measurement Information Systems - Short Form (PROMIS-SF). Total scores range from 8 to 40. Higher scores indicate greater maternal sleep disturbances. Data will be analyzed using the total subscale score.
Changes in maternal anger | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Symptoms of anger will be assessed using the anger subscale on the Patient Reported Outcomes Measurement Information Systems - Short Form (PROMIS-SF). Scores range from 5 to 25. Higher scores on this subscale suggest higher levels of anger. Data will be analyzed using the total subscale score.
Change in maternal self-efficacy | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2;11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Maternal self-efficacy will be assessed using the Perceived Maternal Parenting Self-Efficacy (PMP SE) scale, which measures mothers' perceptions on their abilities as a parent. Higher scores indicate a higher degree of maternal self-efficacy. Data will be analyzed using the total PMP SE score.
Change in maternal substance use | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Problematic maternal alcohol use will be assessed using the Alcohol Use Disorder Identification Test, while problematic cannabis use will be examined with the Cannabis use Disorder Identification Test - Revised. Scores on the Alcohol Use Disorder Identification Test range from 0 to 40, and the scores on the Cannabis use Disorder Identification Test - Revised range from 0 to 32. Higher scores on each test suggests more problematic alcohol and/or cannabis use, respectively. Data will be analyzed using total test scores and clinical cut-offs (≥ 8).
Change in maternal substance use motives | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Maternal substance use motives will be assessed using three coping subscales (i.e., coping with anxiety, depression, and boredom) from the Substance Use Motives Measure. Higher cumulative subscale scores indicate greater motive endorsement. Data will be analyzed using the total subscale scores. There are 3 subscales, anxiety coping, depression coping and boredom coping. For the total score, scores range from 12 to 60.
Change in relationship quality | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Relationship quality will be assessed using the Couples Satisfaction Index - 4 Item which assesses how satisfied mothers are in their current relationship. Higher scores indicate higher levels of relationship satisfaction. Scores on the Couples Satisfaction Index - 4 Item range from 0-21. Data will be analyzed using the total scale score.
Change in child temperament | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention).
  Child temperament will be assessed using the effortful control subscale from the Infant Behavior Questionnaire - Very Short - Revised. Scores on this subscale range from 12 to 84. Higher scores indicate more concerning infant behaviour. Data will be analyzed using the total scale score.
Change in child quality of life | To be assessed pre-intervention (T1; up to 2 months before the start of the intervention), immediately after the intervention (T2; 11 weeks after start of intervention), and at a 6-month follow-up (T3).
  Child quality of life will be measured using the The Pediatric Quality of Life Inventory (infant scales). Higher scores indicate better health related quality of life. Scores range from 0 to 100. Data will be analyzed using the total scale score.

OTHER OUTCOMES:
Usability of the BEAM program | To be assessed immediately after the intervention (T2; 11 weeks after start of intervention).
  The mHealth App Usability Questionnaire will be used to assess participant perceptions of the BEAM app. A total score is created, determining how usable participants found the app.
Program engagement | To be assessed immediately after the intervention (T2; 11 weeks after start of intervention).
  Measures of program engagement will be gathered through Google Analytics and back-end app data will be used to assess recommended mHealth engagement variables such as number of logins to the BEAM app, number of forum posts, time spent on the BEAM app, number of videos watched, time spent watching videos, and number of days between first and last engagement with the app. Weekly telehealth group session attendance (yes/no) will be compiled by the clinical team. Analytics and group attendance data will be used to assess retention (number of weeks completed) and completion (participating in >50% of program weeks either via logging onto the BEAM app or attending the weekly group telehealth session).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E Roos, PhD, Principal Investigator — University of Manitoba; Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (e.g. standardized questionnaire responses, aggregated program use data, sociodemographics linked to an identifier number) may be made available on public data platforms such as open science framework or a requirement by a granting agency or journal.
Supporting Information: Study Protocol
Time Frame: Data is expected to be available in early 2024.

REFERENCES:
- [Derived] Joyce KM, Rioux C, MacKinnon AL, Katz LY, Reynolds K, Kelly LE, Klassen T, Afifi TO, Mushquash AR, Clement FM, Chartier M, Xie EB, Penner KE, Hunter S, Berard L, Tomfohr-Madsen L, Roos LE. The Building Emotional Awareness and Mental health (BEAM) program developed with a community partner for mothers of infants: protocol for a feasibility randomized controlled trial. Pilot Feasibility Stud. 2023 Mar 9;9(1):35. doi: 10.1186/s40814-023-01260-y. PMID 36895006